CLINICAL TRIAL: NCT00981123
Title: Non-interventional Study to Observe Efficacy and Usage of Quetiapine in Acute Episodes of Schizophrenia and as Maintenance Therapy Following Standard Clinical Practice in Croatia
Brief Title: Non-interventional (NI) Study to Observe Efficacy and Usage of Quetiapine in Acute Episodes of Schizophrenia and as Maintenance Therapy Following Standard Clinical Practice in Croatia
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-NHR-SER-2009/1
Record Dates: First submitted 2009-09-14; First posted 2009-09-22 (Estimated); Last update posted 2011-01-10 (Estimated); Status verified 2011-01

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1

SUMMARY:
Observational, non-comparative, epidemiological study to collect and analyse real life data on schizophrenic patients receiving quetiapine according to the standard medical practice in Croatia. The main objectives are to assess after 6 months of quetiapine therapy severity of illness and global improvement in patients using Clinical Global Impression (CGI) scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients with diagnosis of schizophrenia
* Patients who are already treated with quetiapine for at least 12 weeks (outpatients or hospitalised patients)
* Patients capable of signing ICF

Exclusion Criteria:

* Patients with hypersensitivity to active substance or any of the excipients of this product
* Patients with contraindication for quetiapine therapy according to the approved SmPC

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Outpatients or hospitalised patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
To assess severity of illness and global improvement in patients after 6 months of quetiapine therapy using Clinical Global Impression (CGI) scale | CGI - 2 measures (after 3 and after 6 months of quetiapine therapy)

SECONDARY OUTCOMES:
To measure therapeutic response in schizophrenic patients using BPRS scale | BPRS - 2 measures (after 3 and after 6 months of quetiapine therapy)
To evaluate compliance with the prescribed antipsychotic treatment | CGI - 2 measures (after 3 and after 6 months of quetiapine therapy)
To evaluate prescribing practices for quetiapine in the treatment of schizophrenia in Croatia | 3 measures (at the time of quetiapine therapy introduction, after 3 and 6 m of quetiapine therapy)
To evaluate type and frequency of concomitant therapy | At visit 1 ( day 0) and visit 2 (day 90) recorded all changes in concomitant therapy
To evaluate average number of hospitalisations | At visit 1 ( day 0) and visit 2 (day 90) recorded all changes in numbers of hospitalisations
To evaluate frequency of mental illnesses in patient's family | at visit 1 (day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Marija Gjurovic, MD, MSc, Study Director — AstraZeneca Medical Department; Andreja Hasenohrl, DVM, Study Chair — AstraZeneca Medical Department
Locations (18):
- Croatia (18):
  - Research Site, Bjelovar
  - Research Site, Čakovec
  - Research Site, Dubrovnik
  - Research Site, Karlovac
  - Research Site, Osijek
  - Research Site, Popovača
  - Research Site, Pula
  - Research Site, Rijeka
  - Research Site, Sisak
  - Research Site, Slavonski Brod
  - Research Site, Split
  - Research Site, Šibenik
  - Research Site, Varaždin
  - Research Site, Vinkovci
  - Research Site, Vukovar
  - Research Site, Zabok
  - Research Site, Zadar
  - Research Site, Zagreb